CLINICAL TRIAL: NCT04143243
Title: One-day Life Skills Workshop for Veterans With TBI, Pain, and Psychopathology: Evaluating Efficacy and Mechanism of Change
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D3117-R
Record Dates: First submitted 2019-10-25; First posted 2019-10-29 (Actual); Results first posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Traumatic Brain Injury; Chronic Pain; Post Traumatic Stress Disorder; Depression; Anxiety
Keywords: Acceptance and Commitment Therapy; Veterans; polytrauma; traumatic brain injury; chronic pain; Post Traumatic Stress Disorder; depression; Anxiety
MeSH Terms: conditions — Brain Injuries, Traumatic; Chronic Pain; Stress Disorders, Post-Traumatic; Depression; Anxiety Disorders; Multiple Trauma | interventions — Educational Status; Health Resources; Palliative Care

STUDY DESIGN:
Intervention Model Description: ACT plus Education, Resources and Support ('ACT on Life') workshop compared to Education, Resources, & Support only workshop (ERS)
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients will not be told which group they are being allocated to. Follow-up assessments will be administered by anl interviewer blinded to patient assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ACT on Life (Active Comparator): Acceptance and Commitment Therapy plus Education, Resources and Support ('ACT on Life').
  The ACT+ERS intervention will include: 1) Acceptance and Mindfulness Training (2-3 hours); 2) Committed Action Training (2-3 hours) involving helping Veterans clarify what matters most to them and what they want to stand for in life, how they want to behave, and what sorts of strengths and qualities they want to develop; and; 3) Education, Resources, and Support (1 hour).
  Interventions: Behavioral: ACT on Life
- Education, Resources, and Support (Placebo Comparator): Information provided in the ERS workshop was compiled from existing VHA and community resources. Veterans will be educated about 1) symptoms of depression, anxiety and PTSD and how these conditions do and do not impact daily life and functional ability; 2) common difficulties and challenges with reintegration into civilian life; 3) mild TBI, differences between civilian and Veteran TBIs, shared/crossover symptoms (for example, memory and concentration difficulties, sleep disturbance, irritability can be symptoms of depression, PTSD, and mild TBI); 4) chronic pain; how it is often often misinterpreted as on-going damage, leading to fear of physical activities and resulting in increased sedentary behavior and declines in physical functioning; and 5) treatment options and resources. Basic resource counseling will include guidance on the evidence-based treatments available at VHA. Problem solving, relaxation, and deep breathing techniques will be covered
  Interventions: Behavioral: Education, Resources, and Support

INTERVENTIONS:
Behavioral: ACT on Life — 1 day group workshop of ACT plus ERS
  Other Names: ACT plus ERS
  Arms: ACT on Life
Behavioral: Education, Resources, and Support — 1 day group workshop of Education, Resources, and Support
  Other Names: ERS
  Arms: Education, Resources, and Support

SUMMARY:
Mild traumatic brain injury (mTBI) is the signature wound of Veterans returning from the operations in Iraq and Afghanistan (i.e., OIF/OEF/OND), with up to 20 percent experiencing persistent post-concussive symptoms. Among Veterans with mTBI, the majority also experience stress-based psychopathology (e.g., depression, post-traumatic stress disorder, and/or generalized anxiety disorder) and chronic pain. To cope with distress, pain, and other difficulties, Veterans often turn to maladaptive avoidant coping strategies which offer short term relief but exacerbate/maintain mental health problems and have detrimental long-term effects on social, occupational, and community reintegration. Unfortunately, Veterans face important barriers to seeking mental health treatment, including stigma and logistical issues. This proposal aims to examine 1) the impact of a Veteran-centered, non-stigmatizing, 1-day "life skills group workshop" on overall distress and reintegration; and 2) the mechanisms by which this treatment might work as well as possible influences on treatment efficacy.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) is the signature wound of Veterans returning from Operations Iraqi Freedom, Operation Enduring Freedom and Operation New Dawn (OIF/OEF/OND), with up to 20 percent exposed to a mild TBI (mTBI) and experiencing persistent post-concussive symptoms. Among those with a mTBI diagnosis, the majority also suffers from stress-based psychopathology (e.g., depression, post-traumatic stress disorder, generalized anxiety disorder), as well as chronic pain. To cope with distress, pain, and other difficulties, Veterans often turn to maladaptive avoidant coping strategies which offer short term relief but exacerbate/maintain mental health problems and have detrimental long-term effects on social, occupational, and community reintegration. Unfortunately, Veterans face significant barriers to engaging in mental health treatment, including stigma, the belief that one should overcome psychological difficulties on his/her own, and concern that receiving such care would negatively impact their careers. Practical barriers, including time constraints, distance from a treatment facility, and competing priorities (e.g., work and family demands), are also barriers to care. Even among Veterans who start mental health treatment, only a small minority complete a recommended course of evidence-based therapy.

Acceptance and Commitment Therapy (ACT) is a trans-diagnostic treatment model that helps patients to overcome avoidance by promoting acceptance-based coping and engagement in meaningful life activities. In this context, Veterans are asked to think about their "new mission(s)" after leaving the military and the importance of engaging in actions that fulfill their mission even when it may be difficult. ACT has established efficacy in the treatment of depression, anxiety, and chronic pain, and has been effectively implemented in various treatment-delivery formats, including 1-day group workshops. A 1-day ACT workshop addresses specific needs of Veterans with mTBI, stress-based psychopathology, and chronic pain (polytrauma triad) and important barriers to treatment. It 1) is trans-diagnostic (i.e., applies to more than one condition); 2) targets avoidance-based coping; 3) cultivates acceptance-based coping and builds on Veteran's values and goals to motivate them to make difficult decisions; 4) is delivered efficiently and thus more accessible; 5) is less stigmatizing and thus acceptable; and 6) address problems with treatment adherence and completion.

With the support of an RR&D SPiRE pilot grant, the PIs developed a 1-day 'ACT on Life' workshop tailored specifically for the needs of Veterans with mTBI, stress-based psychopathology, and chronic pain. Veterans with this polytrauma were then randomly assigned to the 'ACT on Life' workshop (N=20) or to Treatment as Usual (TAU; N=12). All Veterans attending the 1-day ACT workshop completed it, and relative to TAU, exhibited greater improvements in distress and reintegration at the 3-month follow-up (effect sizes .68 and .47, respectively). Building on these promising preliminary findings, the investigators now propose to conduct a more rigorous randomized controlled trial with 212 Veterans to compare the efficacy of the 1-day ACT workshop to an active treatment comparison (Education, Resources, and Support; ERS) on symptoms of distress and social, occupational, and community reintegration. The investigators will also examine mediators and moderators of treatment response to identify which ACT components are directly responsible for treatment effectiveness and whether treatment benefits are constrained by various personal factors.

Establishing the efficacy of a 1-day ACT workshop for OEF/OEF/OND Veterans with mTBI and multiple coexistent conditions addresses key priorities of VHA RR&D: 1. developing interventions which will improve the psychological health status of Veterans who have specific needs; and 2. enhancing the community, social, and occupational reintegration and functioning of post-deployment Veterans so that they may function more fully in society.

ELIGIBILITY:
Inclusion Criteria:

* OIF/OEF/OND Veteran
* Stress-based psychopathology, as operationalized by a diagnosis of major depressive disorder, generalized anxiety disorder, or PTSD on the M.I.N.I. International Neuropsychiatric interview (M.I.N.I.)
* Deployment-related mild TBI according to the definition of VA/DOD Clinical Practice Guidelines and determined by interview on the Boston Assessment of TBI-Lifetime (BAT-L)
* Pain intensity and level of interference reported to be 5 (moderate) on the Defense and Veterans Pain Rating Scale (DVPRS)

Exclusion Criteria:

* History of bipolar disorder or primary psychotic disorder (e.g., schizophrenia, schizoaffective disorder) on the M.I.N.I.
* A current diagnosis of severe substance use disorder on the M.I.N.I.
* Moderate to severe suicide risk on the suicidality scale on the M.I.N.I.
* History of neurological illness not related to TBI (self-reported and confirmed by Dr. Jorge)
* Severe medical illness (e.g. liver failure, severe coronary artery disease and /or heart failure) posing a new and significant stress burden and requiring intensive treatment (self-reported and confirmed by Dr. Jorge)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2024-08-03 (Actual); Study Completion 2024-08-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lilian N. Dindo, PhD, Principal Investigator — Michael E. DeBakey VA Medical Center, Houston, TX
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: OIF/OEF/OND Veterans with deployment-related mTBI, stress-based psychopathology, and pain (polytrauma clinical triad) were recruited from VAMC, outpatient clinics and Veteran Community Organizations.
Pre-assignment Details: Eligible participants were randomized at their enrollment following phone screening. They were excluded if imminent risk of suicide.
Period: Overall Study
Arm/Group | ACT on Life | Education, Resources, and Support
Started | 90 | 86
Completed | 83 | 77
Not Completed | 7 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ACT on Life | Education, Resources, and Support | Total
Number analyzed (Participants) | 90 | 86 | 176
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 90 | 86 | 176
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.6 (7.8) | 40.7 (7.7) | 40.6 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 77 | 73 | 150
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 24 | 43
  Not Hispanic or Latino | 65 | 55 | 120
  Unknown or Not Reported | 6 | 7 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 28 | 25 | 53
  White | 37 | 30 | 67
  More than one race | 2 | 6 | 8
  Unknown or Not Reported | 21 | 24 | 45
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 90 | 86 | 176
Depression, Anxiety, and Stress Symptoms (DASS-21) -TOTAL Score [Mean (Standard Deviation); unit: units on a scale] — The Depression Anxiety and Stress Scale (DASS-21) measure consists of 21 items that measure current symptoms of depression, anxiety, and stress with a total score. It has been used extensively in clinical trials, including those with military populations. Participants are asked to rate the extent to which they have experienced each state over the past week with a 4-point scale (from 0 = did not apply to me at all to 3 = applied to me very much). For total score, scores are summed and range from 0 to 63. Higher total scores indicate more severe symptoms of depression, anxiety and stress.
  units on a scale | 33.6 (10.5) | 34.9 (12.0) | 34.3 (11.3)
Military to Civilian Questionnaire (M2C-Q) [Mean (Standard Deviation); unit: units on a scale] — The Military to Civilian Questionnaire (M2CQ) is a 16-item self-report measure used to assess the difficulty veterans experience during the post-deployment reintegration process. A total score is calculated by dividing the sum of the item scores by the number of items the veteran completed (excluding those marked "Does not apply").The Min possible score is 0 (if all items are answered as "no difficulty" or "does not apply"). Max possible score is 4 (if all items are answered as "extreme difficulty"). Score: 0 - 64 higher scores indicate greater difficulty with reintegration into civilian life.
  units on a scale | 2.55 (0.62) | 2.53 (0.78) | 2.54 (0.70)
The PTSD Checklist for DSM-5 (PCL-5) [Mean (Standard Deviation); unit: units on a scale] — The PCL-5 is a 20-item self-report questionnaire to assess PTSD based on criteria of the DSM-5. This scale is available from the National Center for PTSD and is extensively used in Veteran populations. Each item is rated on a 5-point scale with anchors from "not at all" to "extremely" indicating how much the participant has been bothered by the PTSD symptoms in the past month. A total symptom severity score can be obtained by summing the scores for a range of scores from 0 to 80. A higher total score demonstrates more severe PTSD symptoms.
  units on a scale | 49.7 (14.2) | 51.9 (15.4) | 50.8 (14.8)
Defense and Veterans Pain Rating Scale (DVPRS)-Severity [Mean (Standard Deviation); unit: units on a scale] — The Defense and Veterans Pain Rating Scale (DVPRS) is a pain assessment tool that assesses severity of pain. It uses a numerical scale ranging from 0 to 10 to assess pain intensity. Minimum Score: 0, representing "No pain". Maximum Score: 10, representing "As bad as pain can be, nothing else matters". It is a reliable and valid instrument developed for use in military populations.
  units on a scale | 6.1 (1.4) | 6.3 (1.5) | 6.2 (1.4)
Acceptance and Action Questionnaire-II (AAQ-II) [Mean (Standard Deviation); unit: units on a scale] — The AAQ-II is an ACT-specific self-report measure of psychological inflexibility. Seven items are rated on a 7-point scale, ranging from 1 ("never true") to 7 ("always true"), with higher scores reflecting greater levels of psychological inflexibility. The total score is calculated by summing the ratings for each of the seven items. The minimum possible score is 7 (7 items x 1 point each).The maximum possible score is 49 (7 items x 7 points each).
  units on a scale | 33.8 (9.1) | 33.3 (9.5) | 33.5 (9.3)
Valued Living Questionnaire (VLQ)-Success [Mean (Standard Deviation); unit: units on a scale] — VLQ is a self-report measure that assesses engagement in valued areas of life. Participants first rate the importance of 10 life domains. They then rate the degree to which their actions over the past week were consistent with each value, from 1 (not at all consistent) to 10 (extremely consistent). The "success" score is the VLQ Composite Score (range from 10-100) and measures how consistently a person is living in accordance with their stated personal values. A higher score indicates greater alignment between actions and values, which is associated with positive psychological outcomes.
  units on a scale | 50.0 (21.7) | 52.1 (20.9) | 51.0 (21.3)

OUTCOME MEASURES:

1. Primary Outcome: The Depression Anxiety and Stress Scale (DASS-21) -TOTAL Score
Description: The Depression Anxiety and Stress Scale (DASS-21) measure consists of 21 items that measure current symptoms of depression, anxiety, and stress with a total score. It has been used extensively in clinical trials, including those with military populations. Participants are asked to rate the extent to which they have experienced each state over the past week with a 4-point scale (from 0 = did not apply to me at all to 3 = applied to me very much). For total score, scores are summed and range from 0 to 63. Higher total scores indicate more severe symptoms of depression, anxiety and stress.
Time Frame: Through study completion, an average of 6 months following workshop/intervention attendance.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- ACT on Life: Acceptance and Commitment Therapy plus Education, Resources and Support ('ACT on Life').
  The ACT+ERS intervention will include: 1) Acceptance and Mindfulness Training (2-3 hours); 2) Committed Action Training (2-3 hours) involving helping Veterans clarify what matters most to them and what they want to stand for in life, how they want to behave, and what sorts of strengths and qualities they want to develop; and; 3) Education, Resources, and Support (1 hour).
  ACT on Life: 1 day group workshop of ACT plus ERS
Arm/Group | ACT on Life | Education, Resources, and Support
Number analyzed (Participants) | 90 | 86
units on a scale | 28.97 (1.34) | 30.77 (1.38)

2. Primary Outcome: Military to Civilian Questionnaire (M2C-Q)
Description: The Military to Civilian Questionnaire (M2CQ) is a 16-item self-report measure used to assess the difficulty veterans experience during the post-deployment reintegration process. A total score is calculated by dividing the sum of the item scores by the number of items the veteran completed (excluding those marked "Does not apply").The Minimum possible score is 0 (if all items are answered as "no difficulty" or "does not apply"). Maximum possible score is 4 (if all items are answered as "extreme difficulty"). Higher scores on the M2CQ indicate greater difficulty with reintegration into civilian life.
Time Frame: Through study completion, an average of 6 months following workshop/intervention attendance.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | ACT on Life | Education, Resources, and Support
Number analyzed (Participants) | 90 | 86
units on a scale | 2.296 (0.096) | 2.395 (0.099)

3. Secondary Outcome: The PTSD Checklist for DSM-5 (PCL-5)
Description: The PCL-5 is a 20-item self-report questionnaire to assess post-traumatic stress disorder (PTSD) based on criteria of the Diagnostic and Statistical Manual for Mental Disorders - Version 5 (DSM-5). This scale is available from the National Center for PTSD and is extensively used in Veteran populations. Each item is rated on a 5-point scale with anchors from "not at all" to "extremely" indicating how much the participant has been bothered by the PTSD symptoms in the past month. A total symptom severity score can be obtained by summing the scores for a range of scores from 0 to 80. A higher total score demonstrates more severe PTSD symptoms.
Time Frame: Through study completion, an average of 6 months following workshop/intervention attendance.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | ACT on Life | Education, Resources, and Support
Number analyzed (Participants) | 90 | 86
units on a scale | 42.38 (1.94) | 47.36 (1.99)

4. Secondary Outcome: Defense and Veterans Pain Rating Scale (Pain Severity)
Description: The Defense and Veterans Pain Rating Scale (DVPRS) is a pain assessment tool that assesses severity of pain. It uses a numerical scale ranging from 0 to 10 to assess pain intensity. Minimum Score: 0, representing "No pain". Maximum Score: 10, representing "As bad as pain can be, nothing else matters". It is a reliable and valid instrument developed for use in military populations.
Time Frame: Through study completion, an average of 6 months following workshop/intervention attendance.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | ACT on Life | Education, Resources, and Support
Number analyzed (Participants) | 90 | 86
units on a scale | 5.77 (0.20) | 5.87 (0.21)

5. Other Pre Specified Outcome: Acceptance and Action Questionnaire-II
Description: The Acceptance and Action Questionnaire-II (AAQ-II) is an ACT-specific self-report measure of psychological inflexibility. The AAQ was designed to measure mechanisms hypothesized to be at work in ACT treatments and has been found to mediate behavioral outcomes in ACT interventions. Seven items are rated on a 7-point scale, ranging from 1 ("never true") to 7 ("always true"), with higher scores reflecting greater levels of psychological inflexibility. The total score is calculated by summing the ratings for each of the seven items. The minimum possible score is 7 (7 items x 1 point each).The maximum possible score is 49 (7 items x 7 points each).
  Higher total scores indicate greater levels of psychological inflexibility and experiential avoidance.
Time Frame: Through study completion, an average of 6 months following workshop/intervention attendance.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | ACT on Life | Education, Resources, and Support
Number analyzed (Participants) | 90 | 86
units on a scale | 30.10 (1.18) | 30.78 (1.23)

6. Other Pre Specified Outcome: Valued Living Questionnaire (VLQ) - Success
Description: Valued Living Questionnaire (VLQ) is a self-report measure that assesses engagement in valued areas of life. Participants first rate the importance of 10 life domains (e.g., family, work, friends etc.) on a 10-point Likert scale (1 = not at all important to 10 = extremely important). They then rate the degree to which their actions over the past week were consistent with each value, from 1 (not at all consistent) to 10 (extremely consistent). The "success" score is the VLQ Composite Score and refers to the composite score that measures how consistently a person is living in accordance with their stated personal values. The Valued Living composite is calculated by multiplying the Importance and Consistency responses for each domain and then calculating the mean of those scores. The resulting Valued Living Composite scores can range from 10-100. A higher score indicates greater alignment between actions and values, which is associated with positive psychological outcomes.
Time Frame: Through study completion, an average of 6 months following workshop/intervention attendance.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | ACT on Life | Education, Resources, and Support
Number analyzed (Participants) | 90 | 86
units on a scale | 48.80 (2.38) | 51.54 (2.41)

7. Other Pre Specified Outcome: Self-reported Service Utilization (Emotional Problems)
Description: The outcome measure is either Yes or No and then we computed the percentage of study participants that responded 'yes' on having utilized services for emotional problems from any of the following, medical provider, spiritual provider(priest/minister), psychiatric help or had hospital admission(in or outpatient) or ER admission.
Time Frame: Through study completion, an average of 6 months following workshop/intervention attendance.
Measure: Count of Participants; unit: Participants
Arm/Group | ACT on Life | Education, Resources, and Support
Number analyzed (Participants) | 90 | 86
Participants | 54 | 44

ADVERSE EVENTS:
Time Frame: Through study completion, up to 6 months following workshop attendance.
Description: This is a low-risk study. The investigators are simply providing a workshop to Veterans to teach them more about their difficulties and new ways they may cope. However, if at any time during the study we obtained information about significant and imminent suicidality, we would follow-up by doing a suicide risk assessment and making immediate referrals.
Arm/Group | ACT on Life | Education, Resources, and Support
All-Cause Mortality (participants affected / at risk) | 0/90 | 0/86
Serious Adverse Events (participants affected / at risk) | 0/90 | 0/86
Other Adverse Events (participants affected / at risk) | 2/90 | 2/86
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ACT on Life (N=90) | Education, Resources, and Support (N=86)
Suicidal Ideation (Psychiatric disorders) | 2 | 2 — When suicidal Ideation was reported to study personnel, suicide risk assessment was completed and immediate referrals were made.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-22): https://cdn.clinicaltrials.gov/large-docs/43/NCT04143243/Prot_SAP_001.pdf
  • Informed Consent Form (2020-08-14): https://cdn.clinicaltrials.gov/large-docs/43/NCT04143243/ICF_000.pdf